CLINICAL TRIAL: NCT03301051
Title: A Randomized, Observer-blind, Placebo-controlled, Multicenter, Phase 3 Study to Assess the Efficacy, Safety, and Immunogenicity of a Plant-Derived Quadrivalent Virus-Like Particles Influenza Vaccine in Adults 18-64 Years of Age
Brief Title: Efficacy, Safety, and Immunogenicity of a Plant-Derived Quadrivalent Virus-Like Particles (VLPs) Influenza Vaccine in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medicago (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CP-PRO-QVLP-012
Record Dates: First submitted 2017-09-21; First posted 2017-10-04 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Virus Diseases; RNA Virus Infections; Respiratory Tract Diseases; Respiratory Tract Infections; Influenza
Keywords: Influenza; Human; RNA Virus Infections; Efficacy; Immunologic; Immunogenic Factors; Physiological Effects of Drug; Virus Diseases; Orthomyxoviridae Infections; Infection; Vaccine; Safety; Plant-made; Virus-like Particle; Hemagglutinin; Quadrivalent Influenza Vaccine
MeSH Terms: conditions — Virus Diseases; RNA Virus Infections; Respiratory Tract Diseases; Respiratory Tract Infections; Influenza, Human; Orthomyxoviridae Infections; Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Quadrivalent VLP Vaccine (Experimental): Participants received one intramuscular (IM) injection of 0.5 mL of 30 μg/strain of the Quadrivalent VLP Influenza Vaccine on Day 0.
  Interventions: Biological: Quadrivalent VLP Vaccine
- Placebo (Placebo Comparator): Participants received one IM injection of 0.5 mL of placebo on Day 0.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Quadrivalent VLP Vaccine — Single dose of a 30 µg/strain of Quadrivalent VLP Vaccine
  Arms: Quadrivalent VLP Vaccine
Biological: Placebo — Single dose of a Placebo
  Arms: Placebo

SUMMARY:
This Phase 3 study is intended to assess the efficacy of the Quadrivalent VLP Influenza Vaccine during the 2017-2018 influenza season in healthy adults 18 to 64 years of age. One dose of Quadrivalent VLP Influenza Vaccine (30 μg/strain) or of placebo will be administered to approximately 10,000 participants

DETAILED DESCRIPTION:
This randomized, observer-blind, placebo-controlled multicenter, Phase 3 study will be conducted at multiple sites. The composition of the Quadrivalent VLP Influenza Vaccine to be used in this study includes a mix of recombinant H1, H3, and two B hemagglutinin proteins expressed as VLPs for the 2017-2018 influenza virus strains.

Approximately 10,000 healthy male and female participants aged 18 to 64 years will be randomized in a 1:1 ratio into one of two parallel treatment groups, such that approximately 5,000 participants will receive the Quadrivalent VLP Influenza Vaccine at a dose of 30 μg/strain and approximately 5,000 participants will receive the placebo. Within the two treatment groups, participants will be stratified by site and two age groups (18-49 years of age and 50-64 years of age in a 1:1 ratio).

Participants will participate in this study for approximately eight to ten months, during which a first visit will be scheduled on Day 0 for screening and vaccine administration.

ELIGIBILITY:
Inclusion Criteria

Participants must meet all of the following inclusion criteria to be eligible for participation in this study; no protocol waivers are allowed:

1. Participants must have a body mass index (BMI) below 40 kg/m^2;
2. Participants are considered by the Investigator to be reliable and likely to cooperate with the assessment procedures and be available for the duration of the study;
3. Participants must be in good general health prior to study participation, with no clinically relevant abnormalities that could jeopardize participant safety or interfere with study assessments, as assessed by the Principal Investigator or sub-Investigator (thereafter referred as Investigator) and determined by medical history, physical examination, and vital signs; Note: Participants with a pre-existing chronic disease will be allowed to participate if the disease is stable and, according to the Investigator's judgment, the condition is unlikely to confound the results of the study or pose additional risk to the participant by participating in the study. Stable disease is generally defined as no new onset or exacerbation of pre-existing chronic disease three months prior to vaccination. Based on the Investigator's judgment, a participant with more recent stabilization of a disease could also be eligible.
4. Female participants must have a negative urine pregnancy test result at the Screening/Vaccination visit (Visit 1).
5. Female participants of childbearing potential must use an effective method of contraception for one month prior to vaccination and agree to continue employing adequate birth control measures for at least 60 days post-vaccination. Moreover, female participants must have no plan to become pregnant for at least two months post-vaccination. Abstinent participants should be asked what method(s) they would use should their circumstances change, and participants without a well-defined plan should be excluded. The following relationship or methods of contraception are considered to be effective:

   * Hormonal contraceptives (e.g. oral, injectable, topical [patch], or estrogenic vaginal ring);
   * Intra-uterine device with or without hormonal release;
   * Male partner using a condom plus spermicide or sterilized partner (at least one year prior to vaccination);
   * Credible self-reported history of heterosexual vaginal intercourse abstinence until at least 60 days post-vaccination;
   * Female partner;
6. Non-childbearing females are defined as:

   * Surgically-sterile (defined as bilateral tubal ligation, hysterectomy or bilateral oophorectomy performed more than one month prior to vaccination); or
   * Post-menopausal (absence of menses for 24 consecutive months and age consistent with natural cessation of ovulation).

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from participating in this study; no protocol waivers are allowed:

1. Any participant whose medical condition(s) is sufficiently severe that annual influenza vaccination would be routinely recommended in the jurisdiction of recruitment, as per the Investigator's judgement;
2. According to the Investigator's opinion, history of significant acute or chronic, uncontrolled medical or neuropsychiatric illness. 'Uncontrolled' is defined as:

   * Requiring a new medical or surgical treatment during the three months prior to study vaccine administration unless the criteria outlined in inclusion criterion no. 5 can be met (i.e. the Investigator can justify inclusion based upon the innocuous nature of medical/surgical events and/or treatments);
   * Requiring any significant change in a chronic medication (i.e. drug, dose, frequency) during the three months prior to study vaccine administration due to uncontrolled symptoms or drug toxicity unless the innocuous nature of the medication change meets the criteria outlined in inclusion criterion no. 5 and is appropriately justified by the Investigator.
3. Any medical or neuropsychiatric condition or any history of excessive alcohol use or drug abuse which, in the Investigator's opinion, would render the participant unable to provide informed consent or unable to provide valid safety observations and reporting;
4. Any autoimmune disease other than hypothyroidism on stable replacement therapy (including, but not limited to rheumatoid arthritis, systemic lupus erythematosus, Crohn's disease, and inflammatory bowel disease) or any confirmed or suspected immunosuppressive condition or immunodeficiency including known or suspected human immunodeficiency virus (HIV), Hepatitis B or C infection, the presence of lymphoproliferative disease;
5. History of chronic pulmonary (including asthma, bronchopulmonary dysplasia, and cystic fibrosis) or cardiovascular (except isolated hypertension), renal, hepatic, neurologic, hematologic (including anemia and hemoglobinopathy), or metabolic disorders (including diabetes mellitus);
6. Because this is a placebo-controlled study, any participants in close contact with individuals considered to be at high risk for developing influenza-related complications (individuals considered at high risk for complications include adults and children who have chronic pulmonary or cardiovascular [except isolated hypertension], renal, hepatic, neurologic, hematologic, or metabolic disorders [including diabetes mellitus]).
7. Administration or planned administration of any non-influenza vaccine within 30 days prior to randomization up to blood sampling on Day 21. Immunization on an emergency basis will be evaluated case-by-case by the Investigator;
8. Administration of any adjuvanted or investigational influenza vaccine within one year prior to randomization or planned administration prior to the completion of the study;
9. Administration of any 'standard', non-adjuvanted influenza vaccine (e.g. live attenuated trivalent/quadrivalent inactivated influenza vaccine or split trivalent/quadrivalent inactivated influenza vaccine administered by intranasal, intradermal, or intramuscular route) within six months prior to randomization and up to completion of the study;
10. Use of any investigational or non-registered product within 30 days or five half-lives, whichever is longer, prior to randomization or planned use during the study period. Participants may not participate in any other investigational or marketed drug study while participating in this study until after the study;
11. Treatment with systemic glucocorticoids at a dose exceeding 10 mg of prednisone (or equivalent) per day for more than seven consecutive days or for 10 or more days in total, within one month of study vaccine administration; any other cytotoxic or immunosuppressant drug, or any immunoglobulin preparation within three months of vaccination and until the completion of the study. Low doses of nasal or inhaled glucocorticoids are allowed. Topical steroids are permitted;
12. Any significant disorder of coagulation including, but not limited to, treatment with warfarin derivatives or heparin. Persons receiving prophylactic anti-platelet medications (e.g. low-dose aspirin [no more than 325 mg/day]), and without a clinically apparent bleeding tendency are eligible. Participants treated with new generation drugs that do not increase the risk of intramuscular bleeding (e.g. clopidogrel) are also eligible;
13. History of allergy to any of the constituents of the Quadrivalent VLP Influenza Vaccine or tobacco;
14. History of anaphylactic allergic reactions to plants or plants components;
15. Use of antihistamines with systemic absorption for more than 14 days in the four weeks prior to vaccination or use of antihistamines 48 hours prior to study vaccination (the use of topical antihistamines and nasal or inhaled steroids is acceptable);
16. Use of prophylactic medications (e.g. acetaminophen/paracetamol, aspirin, naproxen, or ibuprofen) within 24 hours of randomization to prevent or pre-empt symptoms due to vaccination. Any participant discovered to have taken a prophylactic medication to prevent or pre-empt symptoms due to vaccination within the 24 hours prior to planned randomization must be delayed until at least the 24 hours period is met;
17. Planned use of influenza antiviral treatment medication before the collection of nasopharyngeal swabs (e.g. oseltamivir, zanamivir, rapivab);
18. Have a rash, dermatological condition, tattoos, muscle mass, or any other abnormalities at the injection site that may interfere with injection site reaction rating;
19. Participants who have received a blood transfusion within 90 days prior to study vaccination;
20. Any female participant who has a positive or doubtful pregnancy test result prior to vaccination or who is lactating;
21. Participants with abnormal vital signs (systolic blood pressure [BP] > 140 mmHg and/or diastolic BP ≥ 90 mmHg, heart rate ≤ 45 beats/min and ≥ 100 beats/min) evaluated by an Investigator to be clinically significant. A participant with abnormal vital signs results may be included in the study based on Investigator's judgment (e.g. a resting hear rate ≤ 45 in highly trained athletes);
22. Presence of any febrile illness (including an oral temperature ≥ 38.0 ˚C within 24 hours prior to vaccination. Such participants may be re-evaluated for enrolment after resolution of illness;
23. Cancer or treatment for cancer within three years prior to study vaccine administration.

    Persons with a history of cancer who are disease-free without treatment for three years or more are eligible. However, individuals with conditions such as treated and uncomplicated basal cell carcinoma of the skin or non-treated, non-disseminated local prostate cancer may be eligible;
24. Participants identified as an Investigator or employee of the Investigator or clinical site with direct involvement in the proposed study, or identified as an immediate family member (i.e. parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study or any employee of Medicago;
25. Participants with a history of Guillain-Barré Syndrome.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10160 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Medicago
Locations (73):
- United States (29):
  - Site 222, Mobile, Alabama
  - Site 210, Anaheim, California
  - Site 223, Milford, Connecticut
  - Site 217, Coral Gables, Florida
  - Site 220, Hollywood, Florida
  - Site 212, South Miami, Florida
  - Site 203, Savannah, Georgia
  - Site 218, Stockbridge, Georgia
  - Site 206, Wichita, Kansas
  - Site 202, Metairie, Louisiana
  - Site 225, St Louis, Missouri
  - Site 224, Norfolk, Nebraska
  - Site 208, Omaha, Nebraska
  - Site 213, Las Vegas, Nevada
  - Site 205, Binghamton, New York
  - Site 228, Endwell, New York
  - Site 216, Charlotte, North Carolina
  - Site 221, Charlotte, North Carolina
  - Site 227, Winston-Salem, North Carolina
  - Site 201, Columbus, Ohio
  - Site 207, Dakota Dunes, South Dakota
  - Site 209, Bristol, Tennessee
  - Site 204, Austin, Texas
  - Site 229, Austin, Texas
  - Site 226, Fort Worth, Texas
  - Site 219, Fort Worth, Texas
  - Site 214, Salt Lake City, Utah
  - Site 211, West Jordan, Utah
  - Site 230, Norfolk, Virginia
- Canada (10):
  - Site 105, Halifax, Nova Scotia
  - Site 106, Truro, Nova Scotia
  - Site 107, Brampton, Ontario
  - Site 110, Greater Sudbury, Ontario
  - Site 108, Toronto, Ontario
  - Site 109, Mirabel, Quebec
  - Site 103, Pierrefonds, Quebec
  - Site 101, Québec, Quebec
  - Site 102, Québec, Quebec
  - Site 104, Sherbrooke, Quebec
- Finland (10):
  - Site 306, Espoo
  - Site 305, Helsinki
  - Site 310, Helsinki
  - Site 304, Jarvenpaa
  - Site 309, Kokkola
  - Site 307, Oulu
  - Site 303, Pori
  - Site 308, Seinäjoki
  - Site 301, Tampere
  - Site 302, Turku
- Germany (6):
  - Site 402, Berlin
  - Site 403, Berlin
  - Site 406, Berlin
  - Site 401, Essen
  - Site 404, Essen
  - Site 405, Hamburg
- Philippines (6):
  - Site 702, City of Muntinlupa
  - Site 704, City of Muntinlupa
  - Site 705, City of Muntinlupa
  - Site 701, Manila
  - Site 703, Manila
  - Site 706, Pasay
- Thailand (7):
  - Site 601, Bangkok
  - Site 603, Bangkok
  - Site 604, Bangkok
  - Site 606, Bangkok
  - Site 607, Bangkok
  - Site 605, Bangkok Noi
  - Site 602, Chiang Mai
- United Kingdom (5):
  - Site 510, Corby
  - Site 507, Gillingham
  - Site 506, Northwood
  - Site 508, Romford
  - Site 509, Shipley

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ward BJ, Makarkov A, Seguin A, Pillet S, Trepanier S, Dhaliwall J, Libman MD, Vesikari T, Landry N. Efficacy, immunogenicity, and safety of a plant-derived, quadrivalent, virus-like particle influenza vaccine in adults (18-64 years) and older adults (>/=65 years): two multicentre, randomised phase 3 trials. Lancet. 2020 Nov 7;396(10261):1491-1503. doi: 10.1016/S0140-6736(20)32014-6. Epub 2020 Oct 13. PMID 33065035

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized in a 1:1 ratio to receive the Quadrivalent virus-like particle (VLP) Influenza Vaccine at a dose of 30 μg/strain or the placebo.
Pre-assignment Details: Participants were healthy adults 18 to 64 years of age assessed during the 2017-2018 influenza season.
Period: Overall Study
Arm/Group | Quadrivalent VLP Vaccine | Placebo
Started | 5077 | 5083
Safety Analysis Set | 5064 | 5072
Vaccinated | 5065 (1 participant randomized to placebo fraudulently received doses at 2 different sites. Placebo (first site) and vaccine (second site).) | 5072
Completed | 4731 | 4711
Not Completed | 346 | 372
Not completed — Adverse Event | 0 | 4
Not completed — Withdrawal by Subject | 59 | 65
Not completed — Lost to Follow-up | 263 | 282
Not completed — Protocol Violation | 1 | 3
Not completed — Physician Decision | 1 | 3
Not completed — Death | 1 | 1
Not completed — Miscellaneous | 8 | 4
Not completed — Randomized, not vaccinated | 13 | 10

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set (SAS) was defined as all participants who received either the Quadrivalent VLP Influenza Vaccine or the placebo.
Groups:
- Quadrivalent VLP Vaccine: Participants received one IM injection of 0.5 mL of 30 μg/strain of the Quadrivalent VLP Influenza Vaccine on Day 0.
- Total: Total of all reporting groups
Arm/Group | Quadrivalent VLP Vaccine | Placebo | Total
Number analyzed (Participants) | 5064 | 5072 | 10136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5064 | 5072 | 10136
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3051 | 3034 | 6085
  Male | 2013 | 2038 | 4051
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 293 | 326 | 619
  Not Hispanic or Latino | 4769 | 4740 | 9509
  Unknown or Not Reported | 2 | 6 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 20 | 18 | 38
  Asian | 1192 | 1185 | 2377
  Native Hawaiian or Other Pacific Islander | 7 | 6 | 13
  Black or African American | 646 | 620 | 1266
  White | 3168 | 3214 | 6382
  More than one race | 23 | 23 | 46
  Unknown or Not Reported | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Occurrences of Protocol-Defined Respiratory Illness Caused by Vaccine-Matched Influenza Strains
Description: Occurrences of protocol-defined respiratory illness caused by vaccine-matched influenza strains were assessed. The vaccine-matched strains included: H1N1 (A/Michigan/45/2015); H3N2 (A/Hong Kong/4801/2014); B/Brisbane (B/Brisbane/60/2008); and B/Phuket (B/Phuket/3073/2013A). The protocol-defined respiratory illness was determined by the occurrence of at least 1 of the following respiratory symptoms: sneezing, stuffy nose, sore throat, cough, sputum production, wheezing, or difficulty breathing. Occurrences of all matched strains are reported.
Time Frame: Day 14 (post-vaccination) up to ~8 months
Population: The Per Protocol (PP) set consisted of the participants who participated in the study until at least the end of the peak period or for at least five months or until the end of the surveillance period.
Measure: Number; unit: Number of cases
Arm/Group | Quadrivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 4814 | 4812
Number of cases | 110 | 169
Statistical Analysis 1: Comparison: Quadrivalent VLP Vaccine vs Placebo; Test type: Other — Vaccine Efficacy (VE) of VLP vaccine versus placebo = (1 - attack rate in vaccinated participants [ARV]/attack rate in unvaccinated participants [ARU]) x 100%; Vaccine Efficacy = 34.9, 95% CI 2-sided [17.6 to 48.6] — The VE success criterion is defined as a >40% lower limit of the two-sided 95% confidence interval (CI)

2. Secondary Outcome: Number of Occurrences of Protocol-Defined Respiratory Illness Cases Caused by Any Laboratory Confirmed Influenza Strain
Description: Occurrences of protocol-defined respiratory illness due to laboratory-confirmed influenza strain (matched, mismatched, and un-typed) were assessed. A protocol-defined respiratory illness was determined by the occurrence of at least 1 of the following respiratory symptoms: sneezing, stuffy nose, sore throat, cough, sputum production, wheezing, or difficulty breathing.
Time Frame: Day 14 (post-vaccination) up to ~8 months
Population: PP Set
Measure: Number; unit: Number of cases
Arm/Group | Quadrivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 4814 | 4812
Number of cases | 213 | 347
Statistical Analysis 1: Comparison: Quadrivalent VLP Vaccine vs Placebo; Test type: Other — VE of VLP vaccine versus placebo = (1 - ARV/ARU) x 100%; Vaccine Efficacy = 38.6, 95% CI 2-sided [27.6 to 48.0] — The VE success criterion is defined as a >40% lower limit of the two-sided 95% CI

3. Secondary Outcome: Number of Occurrences of Laboratory-Confirmed Protocol-Defined Influenza-Like Illness (ILI) Caused by Vaccine-Matched Influenza Strains
Description: Occurrences of protocol-defined ILI due to laboratory-confirmed influenza caused by influenza viral types/subtypes that are matched (and/or antigenically similar) to the strains covered in the vaccine formulation were assessed. A participant is considered to have protocol-defined ILI if the participant met at least one of the following pre-defined respiratory symptoms: sore throat, cough, sputum production, wheezing, or difficulty breathing AND at least one of the following systemic symptoms: fever (defined as a temperature > 37.2 °C or > 99.0 °F), chills, tiredness, headache or myalgia.
Time Frame: Day 14 (post-vaccination) up to ~8 months
Population: PP Set
Measure: Number; unit: Number of cases
Arm/Group | Quadrivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 4814 | 4812
Number of cases | 98 | 148
Statistical Analysis 1: Comparison: Quadrivalent VLP Vaccine vs Placebo; Test type: Other — VE of VLP vaccine versus placebo = (1 - ARV/ARU) x 100%; Vaccine Efficacy = 33.8, 95% CI 2-sided [14.9 to 48.5] — The VE success criterion is defined as a >40% lower limit of the two-sided 95% CI

4. Secondary Outcome: Number of Occurrences of Laboratory-Confirmed ILI Caused by Any Influenza Strain
Description: Occurrences of laboratory-confirmed ILI caused by any influenza viral strains were assessed. A participant is considered to have protocol-defined ILI if the participant met at least one of the following pre-defined respiratory symptoms: sore throat, cough, sputum production, wheezing, or difficulty breathing AND at least one of the following systemic symptoms: fever (defined as a temperature > 37.2 °C or > 99.0 °F), chills, tiredness, headache or myalgia.
Time Frame: Day 14 (post-vaccination) up to ~8 months
Population: PP Set
Measure: Number; unit: Number of cases
Arm/Group | Quadrivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 4814 | 4812
Number of cases | 178 | 285
Statistical Analysis 1: Comparison: Quadrivalent VLP Vaccine vs Placebo; Test type: Other — VE of VLP vaccine versus placebo = (1 - ARV/ARU) x 100%; Vaccine Efficacy = 37.6, 95% CI 2-sided [25.1 to 48.0] — The VE success criterion is defined as a >40% lower limit of the two-sided 95% CI

5. Secondary Outcome: Number of Occurrences of Protocol-Defined ILI Cases
Description: Occurrences of protocol-defined ILI cases (confirmed or not) were assessed. A participant is considered to have protocol-defined ILI if the participant met at least one of the following pre-defined respiratory symptoms: sore throat, cough, sputum production, wheezing, or difficulty breathing AND at least one of the following systemic symptoms: fever (defined as a temperature > 37.2 °C or > 99.0 °F), chills, tiredness, headache or myalgia.
Time Frame: Day 14 (post-vaccination) up to ~8 months
Population: PP Set
Measure: Number; unit: Number of cases
Arm/Group | Quadrivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 4814 | 4812
Number of cases | 1576 | 1679
Statistical Analysis 1: Comparison: Quadrivalent VLP Vaccine vs Placebo; Test type: Other — VE of VLP vaccine versus placebo = (1 - ARV/ARU) x 100%; Vaccine Efficacy = 6.2, 95% CI 2-sided [0.8 to 11.3] — The VE success criterion is defined as a >40% lower limit of the two-sided 95% CI

6. Secondary Outcome: Number of Participants With at Least One Immediate Complaint
Description: Immediate complaints were defined as any solicited local or systemic reactions. Solicited local reactions included: erythema, swelling, and pain at the injection site and solicited systemic reactions included: fever, headache, fatigue, muscle aches, joint aches, chills, a feeling of general discomfort, swelling in the axilla, and swelling in the neck.
Time Frame: 15 minutes post vaccination
Population: SAS
Measure: Number; unit: Participants
Arm/Group | Quadrivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 5064 | 5072
Participants | 441 | 377

7. Secondary Outcome: Number of Participants With at Least One Solicited Local and Systemic Reactions
Description: Participants were monitored for both solicited local reactions (erythema, swelling, and pain at the injection site) and solicited systemic reactions (fever, headache, fatigue, muscle aches, joint aches, chills, a feeling of general discomfort, swelling in the axilla, and swelling in the neck). Any solicited local or systemic immediate complaint was also included.
Time Frame: Day 0 (post-vaccination) up to Day 7
Population: SAS
Measure: Number; unit: Participants
Arm/Group | Quadrivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 5064 | 5072
Participants | 2776 | 1723

8. Secondary Outcome: Number of Participants With ≥ Severe Solicited Local and Systemic Reactions
Description: Participants were monitored for both solicited local reactions (erythema, swelling, and pain at the injection site) and solicited systemic reactions (fever, headache, fatigue, muscle aches, joint aches, chills, a feeling of general discomfort, swelling in the axilla, and swelling in the neck). Any solicited local or systemic immediate complaint was also included. The intensity of the solicited reactions was graded as mild (1)-easily tolerated and does not interfere with usual activity; moderate (2)-interferes with daily activity, but the participant is still able to function; severe (3)-incapacitating and the participant is unable to work or complete usual activity or potentially life threatening; (4)-likely to be life-threatening if not treated in a timely manner, according to the Food and Drug Administration (FDA) Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials.
Time Frame: Day 0 (post-vaccination) up to Day 7
Population: SAS
Measure: Number; unit: Participants
Arm/Group | Quadrivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 5064 | 5072
Participants | 75 | 85

9. Secondary Outcome: Number of Participants With ≥ Severe Related Solicited Reactions
Description: Participants were monitored for both solicited local reactions (erythema, swelling, and pain at the injection site) and solicited systemic reactions (fever, headache, fatigue, muscle aches, joint aches, chills, a feeling of general discomfort, swelling in the axilla, and swelling in the neck). The intensity of the solicited reactions was graded according to the FDA Toxicity Grading Scale: mild (1), moderate (2), severe (3) or potentially life threatening (4). The causal relationship with the study vaccine was assessed as "definitely not related" (clearly not related), "probably not related" (no medical evidence), "possibly related" (reasonable possibility of cause and effect), "probably related" (plausible biologic mechanism and temporal relationship) or "definitely related" (direct cause and effect relationship). The ≥ severe events included "severe" and "potentially life-threatening" and the related category included "possibly related", "probably related", and "definitely related."
Time Frame: Day 0 (post-vaccination) up to Day 7
Population: SAS
Measure: Number; unit: Participants
Arm/Group | Quadrivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 5064 | 5072
Participants | 56 | 62

10. Secondary Outcome: Number of Participants With Unsolicited Treatment-Emergent Adverse Events (TEAEs)
Description: Participants were monitored for unsolicited TEAEs (e.g., nasopharyngitis, upper respiratory tract infection, headache, and oropharyngeal pain). An adverse event (AE) or adverse experience was defined as any untoward medical occurrence in a participant or clinical investigation participant who was administered a pharmaceutical product, with or without a causal relationship with the treatment. An AE can be any favorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to a medicinal product. An AE was considered treatment-emergent if it began on or after the date and time of Study Day 0 vaccination.
Time Frame: Day 0 (post-vaccination) up to Day 21
Population: SAS
Measure: Number; unit: Participants
Arm/Group | Quadrivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 5064 | 5072
Participants | 661 | 639

11. Secondary Outcome: Number of Participants With ≥ Severe Unsolicited TEAEs
Description: The intensity of the unsolicited TEAEs was graded as mild (1)-easily tolerated and does not interfere with usual activity; moderate (2)-interferes with daily activity, but the participant is still able to function; severe (3)-incapacitating and the participant is unable to work or complete usual activity or potentially life threatening; (4)-likely to be life-threatening if not treated in a timely manner, according to the FDA Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials. The ≥ Severe events included severe and potentially life-threatening events. AE and TEAEs are defined in outcome measure #10.
Time Frame: Day 0 (post-vaccination) up to Day 21
Population: SAS
Measure: Number; unit: Participants
Arm/Group | Quadrivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 5064 | 5072
Participants | 13 | 25

12. Secondary Outcome: Number of Participants With ≥ Severe Related Unsolicited Reactions
Description: The intensity of the solicited local and systemic reactions was graded as: mild (1), moderate (2), severe (3) or potentially life threatening (4). The causal relationship with the study vaccine was assessed as "definitely not related" (clearly not related), "probably not related" (no medical evidence), "possibly related" (reasonable possibility of cause and effect), "probably related" (plausible biologic mechanism and temporal relationship) or "definitely related" (direct cause and effect relationship). The ≥ severe events included "severe" and "potentially life-threatening" and the related category included "possibly related", "probably related", and "definitely related." AE and TEAEs are defined in outcome measure #10.
Time Frame: Day 0 (post-vaccination) up to Day 21
Population: SAS
Measure: Number; unit: Participants
Arm/Group | Quadrivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 5064 | 5072
Participants | 4 | 6

13. Secondary Outcome: Number of Participants With an Occurrence of Death
Description: The number of participants in each treatment group with an occurrence of death was assessed.
Time Frame: Day 0 up to ~8 months
Population: SAS
Measure: Number; unit: Participants
Arm/Group | Quadrivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 5064 | 5072
Participants | 1 | 2

14. Secondary Outcome: Number of Participants With at Least One Serious TEAE
Description: A serious adverse event (SAE) is an AE that results in death, is life threatening, results in a persistent or significant disability or incapacity, results in or prolongs an existing hospitalization, is a congenital anomaly or birth defect, or is another important medical event. An SAE was considered treatment-emergent if it was aggravated in severity or frequency following the administration of the study vaccine, up to and including the last visit of the study. AE is defined in outcome measure #10.
Time Frame: Day 0 up to ~8 months
Population: SAS
Measure: Number; unit: Participants
Arm/Group | Quadrivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 5064 | 5072
Participants | 55 | 51

15. Secondary Outcome: Number of Participants With at Least One AE Leading to Withdrawal
Description: An AE or adverse experience was defined as any untoward medical occurrence in a participant or clinical investigation participant who was administered a pharmaceutical product, with or without a causal relationship with the treatment. An AE can be any favorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to a medicinal product. The number of participants with at least one adverse event leading to withdrawal was assessed.
Time Frame: Day 0 up to ~8 months
Population: SAS
Measure: Number; unit: Participants
Arm/Group | Quadrivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 5064 | 5072
Participants | 0 | 5

16. Secondary Outcome: Number of Participants With at Least One New Onset Chronic Diseases (NOCDs)
Description: All NOCDs that may plausibly have an allergic, autoimmune or inflammatory component were assessed and reported. Plausibility should be interpreted broadly; the only clear exceptions are degenerative conditions such as osteoarthritis, age-related physiologic changes and life-style diseases In this context, most cancers, cardiac conditions and kidney diseases should be reported.
Time Frame: Day 0 up to ~8 months
Population: SAS
Measure: Number; unit: Participants
Arm/Group | Quadrivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 5064 | 5072
Participants | 54 | 41

17. Secondary Outcome: Geometric Mean Titers (GMTs) of Hemagglutination Inhibition (HI) Antibody Response for Each Homologous and Heterologous Influenza Strain
Description: The GMTs in each treatment group were measured using a HI assay for the homologous strains: H1 A/Michigan/45/2015 (H1N1), A/Hong Kong/4801/2014 (H3N2), B/Brisbane/60/2008, B/Phuket/3073/2013, and the heterologous strains: A/Brisbane/59/2007 (IVR-148) (HIN1), A/Uruguay/716/2007 (H3N2), B/Florida/4/2006, B/Malaysia/2506/2004.
Time Frame: Day 0 (pre-vaccination), Day 21
Population: Immunogenicity Per Protocol (IPP) Set consisted of a subset of participants who participated in the immunogenicity portion of the study, who had a Day 21 immunogenicity sample collection.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Quadrivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 278 | 97
Titers
  Homologous (HIN1): Day 0 | 24.2 [20.7 to 28.3] | 30.0 [22.9 to 39.3]
  Homologous (HIN1): Day 21 | 84.8 [71.4 to 100.8] | 27.8 [21.6 to 35.9]
  Homologous (H3N2): Day 0 | 26.2 [21.8 to 31.4] | 29.0 [21.9 to 38.4]
  Homologous (H3N2): Day 21 | 144.9 [121.9 to 172.4] | 28.0 [20.9 to 37.4]
  Homologous (B/Brisbane/60/2008): Day 0 | 12.8 [11.3 to 14.4] | 12.9 [10.6 to 15.7]
  Homologous (B/Brisbane/60/2008): Day 21 | 28.1 [24.8 to 31.9] | 12.1 [10.0 to 14.8]
  Homologous (B/Phuket/3073/2013): Day 0 | 28.8 [24.5 to 33.9] | 28.1 [21.7 to 36.5]
  Homologous (B/Phuket/3073/2013): Day 21 | 87.8 [74.3 to 103.9] | 26.4 [20.4 to 34.1]
  Heterologous (HIN1): Day 0 | 14.5 [12.7 to 16.6] | 14.5 [12.0 to 17.5]
  Heterologous (HIN1): Day 21 | 16.4 [14.4 to 18.8] | 14.4 [11.8 to 17.6]
  Heterologous (H3N2): Day 0 | 17.2 [14.7 to 20.2] | 19.7 [15.4 to 25.3]
  Heterologous (H3N2): Day 21 | 44.1 [37.1 to 52.3] | 17.7 [13.9 to 22.6]
  Heterologous (B/Florida/4/2006): Day 0 | 26.8 [22.8 to 31.6] | 31.5 [24.2 to 41.1]
  Heterologous (B/Florida/4/2006): Day 21 | 65.3 [55.8 to 76.5] | 26.0 [20.1 to 33.7]
  Heterologous (B/Malaysia/2506/2004): Day 0 | 11.5 [10.2 to 12.9] | 10.7 [8.8 to 13.0]
  Heterologous (B/Malaysia/2506/2004): Day 21 | 24.6 [21.6 to 27.9] | 10.6 [8.7 to 12.9]

18. Secondary Outcome: Percentage of Participants With Seroconversion Measured by HI Antibody Response for Each Homologous and Heterologous Strain
Description: Seroconversion rate: the percentage of participants in a given treatment group with either a ≥ 4-fold increase in reciprocal HI titers between Day 0 and Day 21 or a rise of undetectable HI titer (i.e. < 10) pre-vaccination (Day 0) to an HI titer of ≥ 40 on Day 21 was measured using an HI assay for the homologous strains: H1 A/Michigan/45/2015 (H1N1), A/Hong Kong/4801/2014 (H3N2), B/Brisbane/60/2008, B/Phuket/3073/2013, and the heterologous strains: A/Brisbane/59/2007 (IVR-148) (HIN1), A/Uruguay/716/2007 (H3N2), B/Florida/4/2006, B/Malaysia/2506/2004.
Time Frame: Day 0 (pre-vaccination) up to Day 21
Population: IPP Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Quadrivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 278 | 97
Percentage of Participants
  Homologous (HIN1) | 37.1 [31.4 to 43.0] | 0 [0 to 0]
  Homologous (H3N2) | 46.4 [40.4 to 52.5] | 0 [0 to 0]
  Homologous (B/Brisbane/60/2008) | 17.6 [13.3 to 22.6] | 0 [0 to 0]
  Homologous (B/Phuket/3073/2013) | 31.7 [26.2 to 37.5] | 0 [0 to 0]
  Heterologous (HIN1) | 2.5 [1.0 to 5.1] | 0 [0 to 0]
  Heterologous (H3N2) | 23.0 [18.2 to 28.4] | 0 [0 to 0]
  Heterologous (B/Florida/4/2006) | 27.0 [21.9 to 32.6] | 0 [0 to 0]
  Heterologous (B/Malaysia/2506/2004) | 18.3 [14.0 to 23.4] | 0 [0 to 0]

19. Secondary Outcome: Percentage of Participants With Seroprotection Measured by HI Antibody Response for Each Homologous and Heterologous Strain
Description: Seroprotection rate: the percentage of participants in a given treatment group attaining a reciprocal HI titer of ≥ 40 on Day 21 (the percentage of vaccine recipients with a serum HI titer of at least 1:40 following vaccination) was measured using an HI assay for the homologous strains: H1 A/Michigan/45/2015 (H1N1), A/Hong Kong/4801/2014 (H3N2), B/Brisbane/60/2008, B/Phuket/3073/2013, and the heterologous strains: A/Brisbane/59/2007 (IVR-148) (HIN1), A/Uruguay/716/2007 (H3N2), B/Florida/4/2006, B/Malaysia/2506/2004.
Time Frame: Day 0 (pre-vaccination) up to Day 21
Population: IPP Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Quadrivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 278 | 97
Percentage of Participants
  Homologous (HIN1): Day 0 | 40.6 [34.8 to 46.7] | 47.4 [37.2 to 57.8]
  Homologous (HIN1): Day 21 | 74.8 [69.3 to 79.8] | 39.2 [29.4 to 49.6]
  Homologous (H3N2): Day 0 | 46.4 [40.4 to 52.5] | 46.4 [36.2 to 56.8]
  Homologous (H3N2): Day 21 | 85.3 [80.5 to 89.2] | 48.5 [38.2 to 58.8]
  Homologous (B/Brisbane/60/2008): Day 0 | 19.4 [14.9 to 24.6] | 20.6 [13.1 to 30.0]
  Homologous (B/Brisbane/60/2008: Day 21 | 41.0 [35.2 to 47.0] | 15.5 [8.9 to 24.2]
  Homologous (B/Phuket/3073/2013): Day 0 | 47.5 [41.5 to 53.5] | 46.4 [36.2 to 56.8]
  Homologous (B/Phuket/3073/2013): Day 21 | 76.3 [70.8 to 81.1] | 43.3 [33.3 to 53.7]
  Heterologous (HIN1): Day 0 | 23.4 [18.5 to 28.8] | 16.5 [9.7 to 25.4]
  Heterologous (HIN1): Day 21 | 27.0 [21.9 to 32.6] | 16.5 [9.7 to 25.4]
  Heterologous (H3N2): Day 0 | 31.3 [25.9 to 37.1] | 34.0 [24.7 to 44.3]
  Heterologous (H3N2): Day 21 | 58.6 [52.6 to 64.5] | 29.9 [21.0 to 40.0]
  Heterologous (B/Florida/4/2006): Day 0 | 46.8 [40.8 to 52.8] | 48.5 [38.2 to 58.8]
  Heterologous (B/Florida/4/2006): Day 21 | 70.9 [65.1 to 76.1] | 46.4 [36.2 to 56.8]
  Heterologous (B/Malaysia/2506/2004): Day 0 | 20.1 [15.6 to 25.3] | 15.5 [8.9 to 24.2]
  Heterologous (B/Malaysia/2506/2004): Day 21 | 43.2 [37.3 to 49.2] | 13.4 [7.3 to 21.8]

20. Secondary Outcome: Geometric Mean Fold Ratio (GMFR) of HI Antibody Response for Each Homologous and Heterologous Strain
Description: GMFR, the geometric mean of the ratio of GMTs (Day 21/Day 0) in each treatment group was measured using an HI assay for the homologous strains: H1 A/Michigan/45/2015 (H1N1), A/Hong Kong/4801/2014 (H3N2), B/Brisbane/60/2008, B/Phuket/3073/2013, and the heterologous strains: A/Brisbane/59/2007 (IVR-148) (HIN1), A/Uruguay/716/2007 (H3N2), B/Florida/4/2006, B/Malaysia/2506/2004.
Time Frame: Day 0 (pre-vaccination), Day 21
Population: IPP Set
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Quadrivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 278 | 97
Ratio
  Homologous (HIN1) | 3.4 [3.0 to 3.9] | 1.0 [0.8 to 1.2]
  Homologous (H3N2) | 5.5 [4.7 to 6.3] | 1.0 [0.8 to 1.3]
  Homologous (B/Brisbane/60/2008) | 2.2 [2.0 to 2.4] | 0.9 [0.8 to 1.1]
  Homologous (B/Phuket/3073/2013) | 3.1 [2.7 to 3.4] | 0.9 [0.8 to 1.1]
  Heterologous (HIN1) | 1.1 [1.1 to 1.2] | 1.0 [0.9 to 1.1]
  Heterologous (H3N2) | 2.5 [2.3 to 2.9] | 0.9 [0.8 to 1.1]
  Heterologous (B/Florida/4/2006) | 2.4 [2.2 to 2.7] | 0.9 [0.7 to 1.0]
  Heterologous (B/Malaysia/2506/2004) | 2.2 [2.0 to 2.4] | 1.0 [0.8 to 1.1]

21. Secondary Outcome: GMTs of Microneutralization (MN) Antibody Response for Each Homologous Strain
Description: The GMTs in each treatment group were measured using an MN assay for homologous strains: H1 A/Michigan/45/2015 (H1N1), A/Hong Kong/4801/2014 (H3N2), B/Brisbane/60/2008, B/Phuket/3073/2013.
Time Frame: Day 0 (pre-vaccination), Day 21
Population: IPP Set
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Quadrivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 278 | 97
Titers
  Homologous (HIN1): Day 0 | 88.1 [76.7 to 101.1] | 112.3 [91.1 to 138.6]
  Homologous (HIN1): Day 21 | 366.1 [316.1 to 424.1] | 135.7 [110.4 to 166.9]
  Homologous (H3N2): Day 0 | 46.7 [41.9 to 52.1] | 62.1 [53.1 to 72.6]
  Homologous (H3N2): Day 21 | 120.3 [108.9 to 132.9] | 67.2 [57.0 to 79.1]
  Homologous (B/Brisbane/60/2008): Day 0 | 15.2 [13.8 to 16.7] | 14.9 [12.9 to 17.3]
  Homologous (B/Brisbane/60/2008): Day 21 | 38.2 [34.3 to 42.7] | 16.0 [13.7 to 18.6]
  Homologous (B/Phuket/3073/2013): Day 0 | 18.2 [16.3 to 20.4] | 18.9 [16.0 to 22.3]
  Homologous (B/Phuket/3073/2013): Day 21 | 52.0 [46.1 to 58.6] | 21.3 [18.0 to 25.2]

22. Secondary Outcome: Percentage of Participants With Seroconversion Measured by MN Antibody Response for Each Homologous Strain
Description: Seroconversion rate: the percentage of participants in a given treatment group with either a ≥ 4-fold increase in reciprocal MN titers between Day 0 and Day 21 or a rise of undetectable MN titer (i.e. 7.1) pre-vaccination (Day 0) to an MN titer of ≥ 28.3 at Day 21 post-vaccination were measured using an MN assay for homologous strains: H1 A/Michigan/45/2015 (H1N1), A/Hong Kong/4801/2014 (H3N2), B/Brisbane/60/2008, B/Phuket/3073/2013.
Time Frame: Day 0 (pre-vaccination) up to Day 21
Population: IPP Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Quadrivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 278 | 97
Percentage of Participants
  Homologous (HIN1) | 41.7 [35.9 to 47.8] | 2.1 [0.3 to 7.3]
  Homologous (H3N2) | 28.1 [22.9 to 33.7] | 0 [0 to 0]
  Homologous (B/Brisbane/60/2008) | 30.6 [25.2 to 36.4] | 0 [0 to 0]
  Homologous (B/Phuket/3073/2013) | 31.3 [25.9 to 37.1] | 1.0 [0.0 to 5.6]

23. Secondary Outcome: GMFR of MN Antibody Response for Each Homologous Strain
Description: GMFR, the geometric mean of the ratio of GMTs (Day 21/Day 0) was measured in each treatment group using an MN assay for the homologous strains: H1 A/Michigan/45/2015 (H1N1), A/Hong Kong/4801/2014 (H3N2), B/Brisbane/60/2008, and B/Phuket/3073/2013.
Time Frame: Day 0 (pre-vaccination), Day 21
Population: IPP Set
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Quadrivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 278 | 97
Ratio
  Homologous (HIN1) | 4.0 [3.6 to 4.6] | 1.3 [1.1 to 1.6]
  Homologous (H3N2) | 2.5 [2.2 to 2.7] | 1.2 [1.1 to 1.5]
  Homologous (B/Brisbane/60/2008) | 2.5 [2.3 to 2.8] | 1.1 [0.9 to 1.2]
  Homologous (B/Phuket/3073/2013) | 2.8 [2.6 to 3.1] | 1.1 [1.0 to 1.3]

24. Secondary Outcome: Geometric Mean Area (GMA) of Single Radial Hemolysis (SRH) Antibody Response for Each Homologous Strain
Description: The GMA in each treatment group were measured using an SRH assay for homologous strains: H1 A/Michigan/45/2015 (H1N1), A/Hong Kong/4801/2014 (H3N2), B/Brisbane/60/2008, B/Phuket/3073/2013. The GMA calculations were performed by taking the anti-log of the mean of the log titer transformations.
Time Frame: Day 0 (pre-vaccination), Day 21
Population: IPP Set
Measure: Geometric Mean (95% Confidence Interval); unit: mm^2
Arm/Group | Quadrivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 278 | 97
mm^2
  Homologous (HIN1): Day 0 | 10.3 [8.7 to 12.1] | 15.4 [12.0 to 19.8]
  Homologous (HIN1): Day 21 | 31.4 [27.6 to 35.7] | 20.9 [16.4 to 26.6]
  Homologous (H3N2): Day 0 | 15.6 [12.9 to 18.8] | 19.3 [14.2 to 26.1]
  Homologous (H3N2): Day 21 | 56.0 [50.2 to 62.5] | 28.4 [21.2 to 38.1]
  Homologous (B/Brisbane/60/2008): Day 0 | 8.2 [6.9 to 9.9] | 6.8 [5.0 to 9.3]
  Homologous (B/Brisbane/60/2008): Day 21 | 31.9 [27.4 to 37.1] | 9.3 [6.7 to 12.9]
  Homologous (B/Phuket/3073/2013): Day 0 | 11.4 [9.5 to 13.7] | 11.7 [8.8 to 15.7]
  Homologous (B/Phuket/3073/2013): Day 21 | 36.7 [31.9 to 42.1] | 15.5 [11.5 to 20.8]

25. Secondary Outcome: Percentage of Participants With Seroconversion Measured by SRH Antibody Response for Each Homologous Strain
Description: Seroconversion rate: the percentage of participants in a given treatment group showing at least 50 % increase in GMA between Days 0 and 21 were measured using a SRH assay for homologous strains: H1 A/Michigan/45/2015 (H1N1), A/Hong Kong/4801/2014 (H3N2), B/Brisbane/60/2008, B/Phuket/3073/2013.
Time Frame: Day 0 (pre-vaccination) up to Day 21
Population: IPP Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Quadrivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 278 | 97
Percentage of Participants
  Homologous (HIN1) | 53.6 [47.5 to 59.6] | 14.4 [8.1 to 23.0]
  Homologous (H3N2) | 48.2 [42.2 to 54.2] | 14.4 [8.1 to 23.0]
  Homologous (B/Brisbane/60/2008) | 45.7 [39.7 to 51.7] | 9.3 [4.3 to 16.9]
  Homologous (B/Phuket/3073/2013) | 47.1 [41.1 to 53.2] | 12.4 [6.6 to 20.6]

26. Secondary Outcome: Percentage of Participants With Seroprotection Measured by SRH Antibody Response for Each Homologous Strain
Description: Seroprotection rate: the percentage of participants in a given treatment group attaining an area ≥ 25 mm^2 following vaccination (Day 21) were measured using an SRH assay for homologous strains: H1 A/Michigan/45/2015 (H1N1), A/Hong Kong/4801/2014 (H3N2), B/Brisbane/60/2008, B/Phuket/3073/2013.
Time Frame: Day 0 (pre-vaccination) up to Day 21
Population: IPP Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Quadrivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 278 | 97
Percentage of Participants
  Homologous (HIN1): Day 0 | 36.3 [30.7 to 42.3] | 42.3 [32.3 to 52.7]
  Homologous (HIN1): Day 21 | 75.9 [70.4 to 80.8] | 57.7 [47.3 to 67.7]
  Homologous (H3N2): Day 0 | 54.7 [48.6 to 60.6] | 57.7 [47.3 to 67.7]
  Homologous (H3N2): Day 21 | 92.1 [88.3 to 95.0] | 74.2 [64.3 to 82.6]
  Homologous (B/Brisbane/60/2008): Day 0 | 40.3 [34.5 to 46.3] | 37.1 [27.5 to 47.5]
  Homologous (B/Brisbane/60/2008): Day 21 | 81.3 [76.2 to 85.7] | 45.4 [35.2 to 55.8]
  Homologous (B/Phuket/3073/2013): Day 0 | 47.5 [41.5 to 53.5] | 44.3 [34.2 to 54.8]
  Homologous (B/Phuket/3073/2013): Day 21 | 81.7 [76.6 to 86.0] | 54.6 [44.2 to 64.8]

27. Secondary Outcome: GMFR of SRH Antibody Response for Each Homologous Strain
Description: GMFR, the geometric mean of the ratio of GMTs (Day 21/Day 0) was measured in each treatment group using an SRH assay for the homologous strains: H1 A/Michigan/45/2015 (H1N1), A/Hong Kong/4801/2014 (H3N2), B/Brisbane/60/2008, and B/Phuket/3073/2013.
Time Frame: Day 0 (pre-vaccination), Day 21
Population: IPP Set
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Quadrivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 278 | 97
Ratio
  Homologous (HIN1) | 2.9 [2.6 to 3.2] | 1.6 [1.3 to 1.9]
  Homologous (H3N2) | 3.5 [3.1 to 3.9] | 1.6 [1.4 to 2.0]
  Homologous (B/Brisbane/60/2008) | 4.0 [3.5 to 4.5] | 1.3 [1.0 to 1.6]
  Homologous (B/Phuket/3073/2013) | 3.2 [2.9 to 3.6] | 1.3 [1.1 to 1.6]

ADVERSE EVENTS:
Time Frame: Day 0 (post-vaccination) up to ~8 months
Description: SAS. The unsolicited serious adverse events (SAEs), unsolicited non-serious adverse events (NSAEs), and all deaths were reported.
Groups:
- Quadrivalent VLP Vaccine: Participants received one IM injection of 0.5 mL of 30 μg/strain of the Quadrivalent VLP Influenza Vaccine or placebo on Day 0.
Arm/Group | Quadrivalent VLP Vaccine | Placebo
All-Cause Mortality (participants affected / at risk) | 1/5064 | 2/5072
Serious Adverse Events (participants affected / at risk) | 55/5064 | 51/5072
Other Adverse Events (participants affected / at risk) | 930/5064 | 918/5072
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quadrivalent VLP Vaccine (N=5064) | Placebo (N=5072)
Abscess limb (Infections and infestations) | 1 (1) | 1 (1)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 2 (2)
Myelitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal stromal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
Borderline personality disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Drug abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral venous disease (Vascular disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Volvulus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Stag horn calculus (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Complication associated with device (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Snake bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quadrivalent VLP Vaccine (N=5064) | Placebo (N=5072)
Abscess limb (Infections and infestations) | 0 (0) | 2 (2)
Abscess of eyelid (Infections and infestations) | 0 (0) | 1 (1)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 3 (3)
Atypical pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 1 (1)
Bacterial vulvovaginitis (Infections and infestations) | 0 (0) | 1 (1)
Balanitis candida (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 13 (13) | 25 (25)
Bullous impetigo (Infections and infestations) | 1 (1) | 0 (0)
Carbuncle (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 4 (4) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 4 (4) | 7 (7)
Conjunctivitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 6 (6) | 2 (2)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 3 (3) | 4 (5)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 10 (10) | 20 (21)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 2 (2)
Gonorrhoea (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 2 (2)
Hordeolum (Infections and infestations) | 2 (2) | 1 (1)
Impetigo (Infections and infestations) | 1 (1) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 8 (8) | 5 (5)
Kidney infection (Infections and infestations) | 1 (1) | 1 (1)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 2 (2) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 3 (4) | 4 (4)
Mastitis (Infections and infestations) | 1 (1) | 1 (1)
Measles (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 56 (57) | 55 (57)
Oral herpes (Infections and infestations) | 6 (7) | 2 (2)
Oral infection (Infections and infestations) | 1 (2) | 0 (0)
Oropharyngeal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 6 (6) | 3 (3)
Paronychia (Infections and infestations) | 3 (3) | 0 (0)
Pericoronitis (Infections and infestations) | 1 (1) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 10 (10) | 11 (12)
Pharyngitis streptococcal (Infections and infestations) | 11 (12) | 7 (7)
Pharyngotonsillitis (Infections and infestations) | 2 (2) | 2 (2)
Pilonidal cyst (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 8 (8) | 11 (12)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 8 (8) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 31 (38) | 27 (32)
Sinusitis (Infections and infestations) | 24 (26) | 18 (18)
Skin candida (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Systemic viral infection (Infections and infestations) | 1 (1) | 3 (3)
Tonsillitis (Infections and infestations) | 8 (8) | 5 (5)
Tooth abscess (Infections and infestations) | 0 (0) | 7 (7)
Tooth infection (Infections and infestations) | 4 (4) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 126 (139) | 117 (126)
Upper respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 12 (14) | 12 (12)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Varicella zoster virus infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 2 (2)
Viral pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Viral sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 5 (5)
Vulvovaginal mycotic infection (Infections and infestations) | 3 (3) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 5 (5)
Allergy to animal (Immune system disorders) | 0 (0) | 1 (1)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2) | 3 (3)
Seasonal allergy (Immune system disorders) | 1 (1) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypogonadism (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 3 (3) | 2 (2)
Thyroid cyst (Endocrine disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Affect lability (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 7 (7)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 3 (3) | 5 (5)
Insomnia (Psychiatric disorders) | 8 (8) | 5 (5)
Major depression (Psychiatric disorders) | 1 (1) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Aphonia (Nervous system disorders) | 1 (1) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 11 (11) | 9 (9)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 113 (132) | 111 (127)
Hyperaesthesia (Nervous system disorders) | 3 (3) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 2 (2)
Intercostal neuralgia (Nervous system disorders) | 2 (2) | 2 (2)
Loss of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 5 (5) | 6 (6)
Muscle contractions involuntary (Nervous system disorders) | 1 (1) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 3 (3) | 1 (1)
Presyncope (Nervous system disorders) | 3 (3) | 1 (1)
Retinal migraine (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 4 (4)
Sensory loss (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 2 (2) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 2 (2)
Corneal opacity (Eye disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 2 (2) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 1 (1) | 0 (0)
Eye paraesthesia (Eye disorders) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 1 (1)
Eye swelling (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 3 (3)
Ocular hyperaemia (Eye disorders) | 0 (0) | 2 (2)
Photokeratitis (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 4 (4) | 5 (8)
Excessive cerumen production (Ear and labyrinth disorders) | 1 (1) | 0 (0)
External ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 4 (4) | 4 (4)
Vertigo positional (Ear and labyrinth disorders) | 2 (2) | 3 (3)
Arrhythmia (Cardiac disorders) | 0 (0) | 2 (3)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac flutter (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 2 (2)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 3 (3) | 1 (1)
Hypertension (Vascular disorders) | 18 (18) | 16 (16)
Hypertensive crisis (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 39 (39) | 41 (43)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (6)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 49 (51) | 28 (29)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 54 (56) | 57 (61)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 7 (7)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 24 (25) | 28 (28)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 5 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 40 (42) | 39 (40)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 26 (27) | 18 (18)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 10 (10) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 2 (2)
Acid peptic disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Coeliac disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3)
Dental caries (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 14 (14) | 20 (22)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 4 (4)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 3 (3) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 5 (5)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 21 (21) | 10 (10)
Noninfective gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 5 (5) | 4 (4)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Uvulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 13 (13) | 9 (9)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cold urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Guttate psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Ingrown hair (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 6 (7)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (19) | 17 (17)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 22 (23) | 18 (18)
Bursa disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Limb mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 3 (3)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 28 (28) | 28 (28)
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (15) | 6 (6)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypertonic bladder (Renal and urinary disorders) | 2 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bartholin's cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 3 (3) | 4 (4)
Genital rash (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menopausal symptoms (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 2 (2) | 1 (2)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Nipple pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Testicular torsion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Axillary pain (General disorders) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 2 (2) | 5 (5)
Chills (General disorders) | 19 (19) | 13 (13)
Cyst (General disorders) | 0 (0) | 1 (1)
Discomfort (General disorders) | 2 (2) | 2 (2)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 28 (32) | 29 (29)
Feeling hot (General disorders) | 1 (1) | 1 (1)
Hangover (General disorders) | 1 (1) | 1 (1)
Inflammation (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 82 (102) | 87 (122)
Injection site bruising (General disorders) | 1 (1) | 1 (1)
Injection site erythema (General disorders) | 3 (3) | 2 (2)
Injection site haematoma (General disorders) | 1 (1) | 1 (1)
Injection site hypersensitivity (General disorders) | 1 (1) | 0 (0)
Injection site hypoaesthesia (General disorders) | 0 (0) | 1 (1)
Injection site inflammation (General disorders) | 1 (1) | 0 (0)
Injection site oedema (General disorders) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 29 (29) | 8 (8)
Injection site pruritus (General disorders) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 1 (1) | 0 (0)
Injection site warmth (General disorders) | 3 (3) | 0 (0)
Injury associated with device (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 5 (5) | 5 (5)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 4 (4) | 3 (3)
Peripheral swelling (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 11 (11) | 13 (14)
Swelling (General disorders) | 3 (3) | 7 (7)
Vaccination site haematoma (General disorders) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood iron decreased (Investigations) | 2 (2) | 0 (0)
Blood magnesium decreased (Investigations) | 1 (1) | 0 (0)
Blood oestrogen decreased (Investigations) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 0 (0) | 1 (1)
Blood pressure diastolic increased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 5 (5) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 1 (2) | 0 (0)
Influenza B virus test positive (Investigations) | 1 (1) | 1 (1)
Progesterone decreased (Investigations) | 0 (0) | 1 (1)
Respiratory rate increased (Investigations) | 0 (0) | 1 (1)
Vitamin B12 decreased (Investigations) | 1 (1) | 0 (0)
Vitamin D decreased (Investigations) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Animal scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Arthropod sting (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 5 (7) | 3 (3)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Foreign body in eye (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 4 (4) | 7 (7)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Mucosal excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 5 (6) | 5 (5)
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Postoperative fever (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 5 (5) | 10 (10)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Superficial injury of eye (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sexual abuse (Social circumstances) | 1 (1) | 0 (0)
Viral tonsilitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngeal paraesthesia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator understands that the information in the protocol is confidential and should not be disclosed, other than to those directly involved in the execution or the ethical review of the study, without prior written authorization from the Sponsor. It is, however, permissible to discuss information contained in the protocol with a participant in order to obtain consent once Institutional Review Board (IRB) approval is obtained.

DOCUMENTS (2):
  • Study Protocol (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/51/NCT03301051/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/51/NCT03301051/SAP_001.pdf